CLINICAL TRIAL: NCT06039046
Title: Inside Liposarcoma Clinical Trials: Patient Experiences Shared While Undergoing Clinical Trials
Brief Title: Investigating Engagement Patterns and Participation Trends Among Liposarcoma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 90761840
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Liposarcoma
Keywords: Liposarcoma
MeSH Terms: conditions — Liposarcoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study seeks to delve into the firsthand experiences of patients diagnosed with liposarcoma who partake in a separate clinical research featuring a specific medical intervention. The primary emphasis will be on meticulously tracking the rates of trial completion and withdrawal among these individuals.

By joining this clinical study, individuals have the unique opportunity to contribute to the betterment of future liposarcoma patients and play an active role in advancing medical research.

ELIGIBILITY:
Inclusion Criteria:

* Patient has self-identified as planning to enroll in a clinical research
* Patient has been diagnosed with liposarcoma
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Patient does not understand, sign, and return consent form
* Inability to perform regular electronic reporting
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with liposarcoma who are actively considering enrolling in an observational clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to participate in a liposarcoma clinical study | 3 months
Rate of patients who remain in liposarcoma clinical study to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen M, Yang J, Zhu L, Zhou C, Zhao H. Primary intrathoracic liposarcoma: a clinicopathologic study and prognostic analysis of 23 cases. J Cardiothorac Surg. 2014 Jul 4;9:119. doi: 10.1186/1749-8090-9-119. PMID 24993036
- [Background] Marino-Enriquez A, Hornick JL, Dal Cin P, Cibas ES, Qian X. Dedifferentiated liposarcoma and pleomorphic liposarcoma: a comparative study of cytomorphology and MDM2/CDK4 expression on fine-needle aspiration. Cancer Cytopathol. 2014 Feb;122(2):128-37. doi: 10.1002/cncy.21362. Epub 2013 Nov 12. PMID 24227706
- [Background] Rossouw DJ, Cinti S, Dickersin GR. Liposarcoma. An ultrastructural study of 15 cases. Am J Clin Pathol. 1986 Jun;85(6):649-67. doi: 10.1093/ajcp/85.6.649. PMID 3706206

DOCUMENTS (1):
  • Informed Consent Form (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT06039046/ICF_000.pdf